CLINICAL TRIAL: NCT01555411
Title: Akershus Cardiac Examination 1950 Study - a Cohort Study on Cardio- and Cerebrovascular Disease in 62-65-year-old Subjects
Brief Title: Akershus Cardiac Examination (ACE) 1950 Study
Acronym: ACE1950
Status: Active, not recruiting | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/1475 C; AFIA (initial study name) (Other: Vestre Viken Hospital Trust and Akershus University Hospital)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Heart Failure; Mild Cognitive Impairment; Cardiovascular Diseases; Cerebrovascular Disorders
Keywords: Cardiovascular epidemiology; Prospective, observational cohort study; Biomarkers; Cardio- and cerebrovascular imaging
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Cognitive Dysfunction; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, including for genetic testing, and urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Akershus Cardiac Examination (ACE) 1950 Study is a large, observational, prospective, longitudinal, population-based cohort study. The overall aim is to establish an extensive cardio- and cerebrovascular age cohort of elderly subjects for various longitudinal long-term follow-up studies of cardiovascular and cerebrovascular disease.

DETAILED DESCRIPTION:
Design: The Akershus Cardiac Examination (ACE) 1950 Study is a population-based, prospective, cerebro- and cardiovascular age-cohort study of all men and women born in 1950 in Akershus County, Norway.

Time schedule: Study inclusion and baseline examinations took place in the period September 2012 - May 2015.

Current status: 10-year follow-up examinations of all participants are undertaken in 2023-2025, and sub-studies are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Resident in Akershus County (as per October 2011, prior to study invitation)
* Born in the year of 1950
* Ability to consent to participation

Ages: 62 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Akershus County, Norway, born in 1950.
Sampling Method: Non-Probability Sample
Enrollment: 3706 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcomes related to CVD and CV-associated conditions | Maximum 35 years

SECONDARY OUTCOMES:
Specific CV endpoints; e.g. acute myocardial infarction, heart failure, atrial fibrillation, etc. | Maximum 35 years
Specific CV-associated conditions, including renal, cerebrovascular, pulmonary, etc. | Maximum 35 years
Specific clinical phenotypes; e.g. myocardial and arterial structure and function, lung function, etc. | Maximum 35 years

OTHER OUTCOMES:
Impact of left atrial size and function measurements by echocardiography on stroke risk in an 62-65-year-old cohort | Within 35 years
Relation between cognitive function and sub-clinical CVD in a 62-65-year-old Norwegian population cohort | Maximum 35 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnljot Tveit, MD, PhD, Study Director — Vestre Viken Hospital Trust, Department of Medical Research; Helge Røsjø, MD, PhD, Study Director — University Hospital, Akershus; Trygve Berge - member of steering committee, MD, Principal Investigator — Vestre Viken Hospital Trust, Department of Medical Research; Kjetil Steine - member of steering committee, MD, PhD, Principal Investigator — University Hospital, Akershus; Torbjørn Omland - member of steering committee, MD, PhD, Principal Investigator — University Hospital, Akershus; Magnus N Lyngbakken - member of steering committee, MD, Principal Investigator — University Hospital, Akershus
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog, Akershus
  - Vestre Viken HT, Baerum Hospital, Department of Medical Research, Sandvika, Akershus

REFERENCES:
- [Background] Berge T, Vigen T, Pervez MO, Ihle-Hansen H, Lyngbakken MN, Omland T, Smith P, Steine K, Rosjo H, Tveit A; ACE 1950 Study Group. Heart and Brain Interactions--the Akershus Cardiac Examination (ACE) 1950 Study Design. Scand Cardiovasc J. 2015;49(6):308-15. doi: 10.3109/14017431.2015.1086813. Epub 2015 Sep 12. PMID 26364744
- [Result] Ihle-Hansen H, Vigen T, Berge T, Einvik G, Aarsland D, Ronning OM, Thommessen B, Rosjo H, Tveit A, Ihle-Hansen H. Montreal Cognitive Assessment in a 63- to 65-year-old Norwegian Cohort from the General Population: Data from the Akershus Cardiac Examination 1950 Study. Dement Geriatr Cogn Dis Extra. 2017 Sep 28;7(3):318-327. doi: 10.1159/000480496. eCollection 2017 Sep-Dec. PMID 29118784
- [Result] Berge T, Brynildsen J, Larssen HKN, Onarheim S, Jenssen GR, Ihle-Hansen H, Christophersen IE, Myrstad M, Rosjo H, Smith P, Tveit A. Systematic screening for atrial fibrillation in a 65-year-old population with risk factors for stroke: data from the Akershus Cardiac Examination 1950 study. Europace. 2018 Nov 1;20(FI_3):f299-f305. doi: 10.1093/europace/eux293. PMID 29095966
- [Result] Berge T, Lyngbakken MN, Ihle-Hansen H, Brynildsen J, Pervez MO, Aagaard EN, Vigen T, Kvisvik B, Christophersen IE, Steine K, Omland T, Smith P, Rosjo H, Tveit A. Prevalence of atrial fibrillation and cardiovascular risk factors in a 63-65 years old general population cohort: the Akershus Cardiac Examination (ACE) 1950 Study. BMJ Open. 2018 Aug 1;8(7):e021704. doi: 10.1136/bmjopen-2018-021704. PMID 30068617
- [Result] Ihle-Hansen H, Vigen T, Ihle-Hansen H, Ronning OM, Berge T, Thommessen B, Lyngbakken MN, Orstad EB, Enger S, Nygard S, Rosjo H, Tveit A. Prevalence of Carotid Plaque in a 63- to 65-Year-Old Norwegian Cohort From the General Population: The ACE (Akershus Cardiac Examination) 1950 Study. J Am Heart Assoc. 2018 May 8;7(10):e008562. doi: 10.1161/JAHA.118.008562. PMID 29739796
- [Result] Chandra A, Rosjo H, Eide IA, Vigen T, Ihle-Hansen H, Orstad EB, Ronning OM, Lyngbakken MN, Berge T, Schmidt EB, Omland T, Tveit A, Svensson M. Plasma marine n-3 polyunsaturated fatty acids and cardiovascular risk factors: data from the ACE 1950 study. Eur J Nutr. 2020 Jun;59(4):1505-1515. doi: 10.1007/s00394-019-02007-3. Epub 2019 May 23. PMID 31123865
- [Result] Vigen T, Ihle-Hansen H, Lyngbakken MN, Berge T, Thommessen B, Ihle-Hansen H, Orstad EB, Enger S, Ariansen I, Rosjo H, Tveit A, Ronning OM. Blood pressure at age 40 predicts carotid atherosclerosis two decades later: data from the Akershus Cardiac Examination 1950 Study. J Hypertens. 2019 Oct;37(10):1982-1990. doi: 10.1097/HJH.0000000000002131. PMID 31116158
- [Result] Ihle-Hansen H, Vigen T, Berge T, Hagberg G, Engedal K, Ronning OM, Thommessen B, Lyngbakken MN, Nygard S, Rosjo H, Tveit A, Ihle-Hansen H. Carotid Atherosclerosis and Cognitive Function in a General Population Aged 63-65 Years: Data from the Akershus Cardiac Examination (ACE) 1950 Study. J Alzheimers Dis. 2019;70(4):1041-1049. doi: 10.3233/JAD-190327. PMID 31306128
- [Result] Aagaard EN, Kvisvik B, Pervez MO, Lyngbakken MN, Berge T, Enger S, Orstad EB, Smith P, Omland T, Tveit A, Rosjo H, Steine K. Left ventricular mechanical dispersion in a general population: Data from the Akershus Cardiac Examination 1950 study. Eur Heart J Cardiovasc Imaging. 2020 Feb 1;21(2):183-190. doi: 10.1093/ehjci/jez210. PMID 31504360
- [Result] Vigen T, Ihle-Hansen H, Lyngbakken MN, Berge T, Thommessen B, Ihle-Hansen H, Orstad EB, Enger S, Rosjo H, Tveit A, Ronning OM. Carotid Atherosclerosis is Associated with Middle Cerebral Artery Pulsatility Index. J Neuroimaging. 2020 Mar;30(2):233-239. doi: 10.1111/jon.12684. Epub 2019 Dec 30. PMID 31889363
- [Result] Ronningen PS, Berge T, Solberg MG, Enger S, Nygard S, Pervez MO, Orstad EB, Kvisvik B, Aagaard EN, Rosjo H, Tveit A, Steine K. Sex differences and higher upper normal limits for left atrial end-systolic volume in individuals in their mid-60s: data from the ACE 1950 Study. Eur Heart J Cardiovasc Imaging. 2020 May 1;21(5):501-507. doi: 10.1093/ehjci/jeaa004. PMID 32031593
- [Result] Lyngbakken MN, Aagaard EN, Kvisvik B, Berge T, Pervez MO, Brynildsen J, Tveit A, Steine K, Rosjo H, Omland T. Cardiac Troponin I and T Are Associated with Left Ventricular Function and Structure: Data from the Akershus Cardiac Examination 1950 Study. Clin Chem. 2020 Apr 1;66(4):567-578. doi: 10.1093/clinchem/hvaa023. PMID 32227098
- [Result] Chandra A, Rosjo H, Svensson M, Vigen T, Ihle-Hansen H, Orstad EB, Ronning OM, Lyngbakken MN, Nygard S, Berge T, Schmidt EB, Omland T, Tveit A, Eide IA. Plasma linoleic acid levels and cardiovascular risk factors: results from the Norwegian ACE 1950 Study. Eur J Clin Nutr. 2020 Dec;74(12):1707-1717. doi: 10.1038/s41430-020-0641-4. Epub 2020 Apr 27. PMID 32341488
- [Result] Chandra A, Lyngbakken MN, Eide IA, Rosjo H, Vigen T, Ihle-Hansen H, Orstad EB, Ronning OM, Berge T, Schmidt EB, Tveit A, Omland T, Svensson M. Plasma Trans Fatty Acid Levels, Cardiovascular Risk Factors and Lifestyle: Results from the Akershus Cardiac Examination 1950 Study. Nutrients. 2020 May 14;12(5):1419. doi: 10.3390/nu12051419. PMID 32423040
- [Result] Lyngbakken MN, Kvisvik B, Aagaard EN, Berge T, Pervez MO, Brynildsen J, Tveit A, Steine K, Rosjo H, Omland T. B-Type Natriuretic Peptide Is Associated with Indices of Left Ventricular Dysfunction in Healthy Subjects from the General Population: The Akershus Cardiac Examination 1950 Study. Clin Chem. 2021 Jan 8;67(1):204-215. doi: 10.1093/clinchem/hvaa257. PMID 33279958
- [Result] Lyngbakken MN, Vigen T, Ihle-Hansen H, Brynildsen J, Berge T, Ronning OM, Tveit A, Rosjo H, Omland T. Cardiac troponin I measured with a very high sensitivity assay predicts subclinical carotid atherosclerosis: The Akershus Cardiac Examination 1950 Study. Clin Biochem. 2021 Jul;93:59-65. doi: 10.1016/j.clinbiochem.2021.04.005. Epub 2021 Apr 20. PMID 33861986
- [Result] Myhre PL, Lyngbakken MN, Berge T, Roysland R, Aagaard EN, Pervez O, Kvisvik B, Brynildsen J, Norseth J, Tveit A, Steine K, Omland T, Rosjo H. Diagnostic Thresholds for Pre-Diabetes Mellitus and Diabetes Mellitus and Subclinical Cardiac Disease in the General Population: Data From the ACE 1950 Study. J Am Heart Assoc. 2021 Jun;10(11):e020447. doi: 10.1161/JAHA.120.020447. Epub 2021 May 17. PMID 33998259
- [Result] Myhre PL, Heck SL, Skranes JB, Prebensen C, Jonassen CM, Berge T, Mecinaj A, Melles W, Einvik G, Ingul CB, Tveit A, Berdal JE, Rosjo H, Lyngbakken MN, Omland T. Cardiac pathology 6 months after hospitalization for COVID-19 and association with the acute disease severity. Am Heart J. 2021 Dec;242:61-70. doi: 10.1016/j.ahj.2021.08.001. Epub 2021 Aug 13. PMID 34400140
- [Result] Caspersen NF, Soyseth V, Lyngbakken MN, Berge T, Ariansen I, Tveit A, Rosjo H, Einvik G. Treatable Traits in Misdiagnosed Chronic Obstructive Pulmonary Disease: Data from the Akershus Cardiac Examination 1950 Study. Chronic Obstr Pulm Dis. 2022 Apr 29;9(2):165-180. doi: 10.15326/jcopdf.2021.0265. PMID 35158418
- [Result] Ronningen PS, Berge T, Solberg MG, Enger S, Pervez MO, Orstad EB, Kvisvik B, Aagaard EN, Lyngbakken MN, Ariansen I, Rosjo H, Steine K, Tveit A. Impact of Blood Pressure in the Early 40s on Left Atrial Volumes in the Mid-60s: Data From the ACE 1950 Study. J Am Heart Assoc. 2022 Jun 7;11(11):e023738. doi: 10.1161/JAHA.121.023738. Epub 2022 May 27. PMID 35621203
- [Result] Aagaard EN, Lyngbakken MN, Kvisvik B, Berge T, Pervez MO, Ariansen I, Tveit A, Steine K, Rosjo H, Omland T. Associations between cardiovascular risk factors, biomarkers, and left ventricular mechanical dispersion: insights from the ACE 1950 Study. Eur Heart J Open. 2022 Feb 12;2(2):oeac006. doi: 10.1093/ehjopen/oeac006. eCollection 2022 Mar. PMID 35919126
- [Result] Lyngbakken MN, Kvisvik B, Berge T, Pervez MO, Aagaard EN, Ariansen I, Omland T, Tveit A, Steine K, Rosjo H. Serial blood pressure measurements, left ventricular remodelling and cardiovascular outcomes. Eur J Clin Invest. 2023 Jan;53(1):e13876. doi: 10.1111/eci.13876. Epub 2022 Sep 24. PMID 36120822
- [Result] Lyngbakken MN, Ronningen PS, Solberg MG, Berge T, Brynildsen J, Aagaard EN, Kvisvik B, Rosjo H, Steine K, Tveit A, Omland T. Prediction of incident atrial fibrillation with cardiac biomarkers and left atrial volumes. Heart. 2023 Feb 14;109(5):356-363. doi: 10.1136/heartjnl-2022-321608. PMID 36261282
- [Result] Walle-Hansen MM, Berge T, Vigen T, Myrstad M, Hagberg G, Ihle-Hansen H, Sandset EC, Thommessen B, Ariansen IKH, Lyngbakken MN, Rosjo H, Ronning OM, Tveit A, Ihle-Hansen H. Systolic blood pressure at age 40 and cognitive function 25 years later: the Akershus Cardiac Examination (ACE) 1950 Study. J Hypertens. 2023 Jan 1;41(1):132-139. doi: 10.1097/HJH.0000000000003312. Epub 2022 Oct 20. PMID 36453656
- [Result] Ihle-Hansen H, Vigen T, Berge T, Walle-Hansen MM, Hagberg G, Ihle-Hansen H, Thommessen B, Ariansen I, Rosjo H, Ronning OM, Tveit A, Lyngbakken M. Carotid Plaque Score for Stroke and Cardiovascular Risk Prediction in a Middle-Aged Cohort From the General Population. J Am Heart Assoc. 2023 Sep 5;12(17):e030739. doi: 10.1161/JAHA.123.030739. Epub 2023 Aug 23. PMID 37609981
- [Derived] Walle-Hansen MM, Hagberg G, Myrstad M, Berge T, Vigen T, Ihle-Hansen H, Thommessen B, Ariansen I, Lyngbakken MN, Rosjo H, Ronning OM, Beyer MK, Tveit A, Ihle-Hansen H. Blood pressure at age 40 and key features of cerebral small vessel disease at age 70: data from the ACE 1950 Study. BMC Cardiovasc Disord. 2025 Oct 9;25(1):724. doi: 10.1186/s12872-025-05140-6. PMID 41068629
- [Derived] Dypvik R, Fjukstad KK, Lydersen S, Berge T, Tveit A, Rosjo H, Omland T, Einvik G, Lyngbakken MN. Associations Between Growth Differentiation Factor 15 and Anxiety and Depression in the General Population: The Akershus Cardiac Examination 1950 Study. Biopsychosoc Sci Med. 2025 Feb-Mar 01;87(2):153-159. doi: 10.1097/PSY.0000000000001365. PMID 39909014
- [Derived] Walle-Hansen MM, Hagberg G, Myrstad M, Berge T, Vigen T, Ihle-Hansen H, Thommessen B, Ariansen I, Lyngbakken MN, Rosjo H, Ronning OM, Tveit A, Ihle-Hansen H. Systolic blood pressure at age 40 and 30-year stroke risk in men and women. Open Heart. 2024 Aug 22;11(2):e002805. doi: 10.1136/openhrt-2024-002805. PMID 39179252
- [Derived] Ihle-Hansen H, Einvik G, Hagberg G, Thommessen B, Ronning OM, Vigen T, Lyngbakken MN, Berge T, Rosjo H, Tveit A, Ihle-Hansen H. Sleep Duration and Cognitive Function: The Akershus Cardiac Examination 1950 Study. Dement Geriatr Cogn Disord. 2024;53(6):338-344. doi: 10.1159/000540273. Epub 2024 Jul 24. PMID 39047714
- See also: Study website — http://www.ace1950.no